CLINICAL TRIAL: NCT06556563
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Optune® (TTFields, 200 kHz) Concomitant With Maintenance Temozolomide and Pembrolizumab Versus Optune® Concomitant With Maintenance Temozolomide and Placebo for the Treatment of Newly Diagnosed Glioblastoma (EF-41/KEYNOTE D58).
Brief Title: EF-41/KEYNOTE D58: Phase 3 Study of Optune Concomitant With Temozolomide Plus Pembrolizumab in Newly Diagnosed Glioblastoma
Acronym: EF-41
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NovoCure GmbH (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF-41; 2024-513550-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma
Keywords: TTFields; Pembrolizumab; Glioblastoma; Tumor Treating Fields; Immunotherapy; Merck Sharp & Dohme LLC; GBM
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; pembrolizumab

STUDY DESIGN:
Intervention Model Description: The participants in the study will be randomized in a ratio of 2:1 in favor of the treatment group to one of the following groups:
  Treatment Group - Optune concomitant with maintenance TMZ and pembrolizumab.
  Control Group - Optune concomitant with maintenance TMZ and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Device: Optune® device; Drug: Temozolomide; Drug: Pembrolizumab
- Control Group (Placebo Comparator)
  Interventions: Device: Optune® device; Drug: Temozolomide; Drug: Placebo

INTERVENTIONS:
Device: Optune® device — Optune® device delivering TTFields therapy at 200 kHz.
  Other Names: TTFields
Drug: Temozolomide — Temozolomide per approved labeling.
Drug: Pembrolizumab — Pembrolizumab dose throughout this study is 200 mg IV Q3W for a maximum of 35 cycles.
  Arms: Treatment Group
Drug: Placebo — Placebo (saline solution) dose throughout this study is 200 mg IV Q3W for a maximum of 35 cycles.
  Arms: Control Group

SUMMARY:
This is a multicenter, two-arm, randomized, double-blind, placebo-controlled study of Optune® (Tumor Treating Fields at 200 kHz) together with maintenance Temozolomide (TMZ) chemotherapy agent and pembrolizumab compared to Optune® together with maintenance TMZ and placebo in newly diagnosed Glioblastoma (GBM) patients. The primary objective of the study is to evaluate the Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative) has provided documented informed consent for the study.
2. Be ≥ 18 years of age on day of providing informed consent.
3. Participant with new diagnosis of GBM according to World Health Organization (WHO) 2021 Classification.
4. Recovered from maximal debulking surgery (gross total resection, partial resection and biopsy-only patients are all acceptable), Gliadel wafers placement at the time of surgical resection is not allowed.
5. Have completed standard adjuvant chemoradiotherapy of radiotherapy (RT) according to local practice (56-64 Gy), and concomitant TMZ chemotherapy.
6. Amenable to treatment with Optune concomitant with maintenance TMZ (150-200 mg/m^2 daily x 5, Q28 days).
7. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 assessed within 7 days before randomization.
8. Stable or decreasing dose of corticosteroids (dexamethasone ≤ 2mg or equivalent) for the last 7 days prior to randomization, if applicable.

Exclusion Criteria:

1. Has received prior therapy with an anti-Programmed Cell Death 1 (PD-1), anti- Programmed Cell Death-Ligand 1(PD-L1), or anti Programmed Cell Death-Ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g.Cytotoxic T-Lymphocyte-Associated protein 4 (CTLA-4), OX 40, CD137).
2. Ongoing requirement for >2 mg dexamethasone (or equivalent), due to intracranial mass effect.
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization.
4. Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first study treatment.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
7. Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
8. Early progressive disease after the end of TMZ/RT. If pseudo progression is suspected, additional imaging studies should be performed to rule out true progression.
9. Infratentorial or leptomeningeal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months
  Overall survival (OS) is defined as the time from randomization to death due to any cause

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) per RANO 2.0 assessed by investigator | 24 months
  PFS is defined as the time interval, in months, between randomization and the first documented disease progression per RANO 2.0 assessed by investigator or death due to any cause, whichever occurs first.
  Note: RANO 2.0 = Modified Radiographic Response Assessment in Neuro-Oncology
Progression-Free Survival (PFS) per RANO 2.0 assessed by investigator | 24 months
  PFS is defined as the time interval, in months, between randomization and the first documented disease progression per RANO 2.0 assessed by investigator or death due to any cause, whichever occurs first.
  Note: RANO 2.0 = Response Assessment in Neuro-Oncology

CONTACTS AND LOCATIONS:
Locations (81):
- United States (30):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Cancer Institute, Palo Alto, California
  - UF Health Neuromedicine, Gainesville, Florida
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - John Theurer Cancer Center/ Hackensack Meridian Health, Hackensack, New Jersey
  - Northwell Health, Lake Success, New York
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center- Montefiore Medical Park, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Sidney Kimmel Comprehensive Cancer Center, Clinical Trials Organization, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The University of Texas, Houston, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
- Nemocnice Na Homolce, Prague, Czechia
- France (5):
  - Centre Hospitalier Universitaire de Lyon, Bron
  - Hopital de la Timone, Marseille
  - Hopital Saint-Louis, Paris
  - Groupe Hospitalier Pitie - Salpetriere, Paris
  - Institut Claudius Regaud, Toulouse
- Germany (3):
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Essen, Essen
  - University Hospital Frankfurt, Frankfurt
- Israel (4):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center- Beilinson Hospital, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Ospedale Bellaria, Bologna
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Ospedale del Mare, Napoli
  - UOC Oncologia Medica 1 Istituto Oncologico Veneto IOV-IRCCS, Padua
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - U.O.C. Immunoterapia Oncologica A.O.U. Senese, Policlinico Santa Maria alle Scotte, Siena
- Japan (10):
  - Kyushu University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Kanazawa University Hospital, Ishikawa
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Kyorin University Hospital, Mitaka
  - Nagoya University Hospital, Nagoya
  - Saitama Medical University International Medical Center, Saitama
  - Tohoku University Hospital, Sendai
  - National Cancer Center Hospital, Tokyo
- Poland (2):
  - Centrum Onkologii, Bydgoszcz
  - Narodowy Instytut Onkologii, Gliwice
- Spain (9):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia de L'Hospitalet (ICO L'Hospitalet), Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politécnic La Fe, Valencia
- Switzerland (3):
  - University Hospital Basel Medical Oncology, Basel
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - University Hospital Zurich, Zurich
- United Kingdom (8):
  - Queen Elizabeth, Birmingham
  - Addenbrooke's Hospital (Cambridge University Hospitals NHS Foundation Trust), Cambridge
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - The Christie Hospital, Manchester
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Marsden, Sutton

IPD SHARING:
Plan to Share IPD: Undecided